CLINICAL TRIAL: NCT01205529
Title: ST-segment Elevation With Procainamide as an ECG Endophenotype of AF
Brief Title: ST-segment Elevation as an AF Endophenotype
Acronym: Proc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dan Roden, Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB # 100800; U19HL065962 (NIH)
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; ST elevation; Genotype
MeSH Terms: conditions — Atrial Fibrillation | interventions — Procainamide

STUDY DESIGN:
Masking Description: All participants and investigators were blinded to the genetic sequencing results at the time of outcome ascertainment
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AF with ST changes on ECG (Other): Those patients with ST segment or J Point elevation on electrocardiogram. Can be on initial screening electrocardiogram or on electrocardiograms during procainamide infusion. These subjects will harbor cardiac sodium channel gene variants.
  Interventions: Drug: Procainamide

INTERVENTIONS:
Drug: Procainamide — One time intravenous infusion of Procainamide administered over 30 minutes. Dosage is calculated as 10mg/kg based on subject's ideal body weight.

SUMMARY:
The purpose of this study is to look for a similarity in people's genes that may help understand which people could benefit from certain drugs for the treatment of atrial fibrillation (AF).

DETAILED DESCRIPTION:
Current drug therapies to suppress AF are incompletely and unpredictably effective and carry significant (albeit generally small) risks of serious adverse effects, including drug-induced long QT syndrome (diLQTS), other forms of proarrhythmia, increased mortality through uncertain mechanisms, and extracardiac toxicity. Identification of clinical and genetic subtypes of AF will permit stratification of therapeutic approaches and thereby facilitate the practice of personalized medicine. Furthermore, limited success of drug therapy and increase in drug toxicity in AF is probably because the arrhythmia represents a final common pathway of multiple initiating mechanisms, including some that are genetically-defined.

Identifying specific intermediate phenotypes ("endophenotypes") associated with defined clinical courses in AF represents a potential method to systematically subtype patients by underlying mechanism and represents a much-needed clinical advance. Clinical endophenotypes that have been studied include atrial fibrillatory rate, prolonged signal-averaged P-wave duration, and biomarker profiles. The endophenotype we will study here is right precordial ST segment elevation, seen not only in Brugada syndrome (BrS) (where it is unmasked by sodium channel blocking drugs) but also commonly in early-onset ('lone') AF and in patients with AF-associated rare variants in genes encoding the cardiac sodium channel α- or β-subunits. Taken together these data suggest the hypothesis to be tested in this study, that variants in multiple genes can culminate in a similar AF-prone substrate by reducing sodium current that can be identified by screening for baseline or manifest right precordial ST segment elevation endophenotype after sodium channel block with intravenous procainamide.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergoing AF ablation at Vanderbilt or MGH

Exclusion Criteria:

* Patients taking membrane active anti-arrhythmic drugs with sodium channel blocking properties (amiodarone, dronedarone, flecainide, propafenone) at the time of the ablation
* Patients with a history of Brugada syndrome or type 1 Brugada ECG pattern on the baseline ECG
* Patients with a history of drug-induced torsades de pointes
* Patients with a known history of hypersensitivity to procainamide, procaine or related drugs
* Patients with a history of systemic lupus erythematosus and myasthenia gravis
* Patients with a history of second degree AV block (Mobitz type II) or third degree AV block
* Women of child-bearing potential unless post-menopausal, surgically sterile, or have a negative pregnancy test day on the day of procedure
* Patients with dual chamber pacemakers or implantable defibrillators requiring ventricular pacing (uninterpretable ECG)
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2010-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawood Darbar, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Atrial Fibrillation With ST Changes on Electrocardiogram: Those patients with ST segment or J Point elevation on electrocardiogram. Can be on initial screening electrocardiogram or on electrocardiograms during procainamide infusion. These subjects will also have SCN5A mutation.
  Procainamide: One time intravenous infusion of Procainamide administered over 30 minutes. Dosage is calculated as 10mg/kg based on subject's ideal body weight.
Period: Overall Study
Arm/Group | Atrial Fibrillation With ST Changes on Electrocardiogram
Started | 161
Completed | 106
Not Completed | 55
Not completed — Procedure Cancelled | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 4
Not completed — Unstable post op | 15
Not completed — No longer met criteria | 30

BASELINE CHARACTERISTICS:
Arm/Group | Atrial Fibrillation With ST Changes on Electrocardiogram
Number analyzed (Participants) | 161
Age, Continuous [Mean (Full Range); unit: years] | 55 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 120
Region of Enrollment [Number; unit: participants]
  United States | 161

OUTCOME MEASURES:

1. Primary Outcome: ST Segment Elevation ≥ 1.5 mm in the Right Precordial Leads (V1-V3), Either at Baseline or Manifested After Sodium Channel Block With Intravenous Procainamide
Description: Number of participants who demonstrated ST-segment elevation >1.5mm in the right precordial leads (V1-V3) either at baseline or after sodium channel block with intravenous procainamide infusion.
Time Frame: During (5, 10, 15, 20, 25, 30 minutes after initiating) or up to 15 minutes after completion of intravenous procainamide infusion
Population: Number of subject who had >/= 1.5mm right precordial ST-segment elevation at baseline or with procainamide administration
Measure: Count of Participants; unit: Participants
Groups:
- Atrial Fibrillation With ST Changes on Electrocardiogram: Those patients with ST segment or J Point elevation on electrocardiogram. Can be on initial screening electrocardiogram or on electrocardiograms during procainamide infusion. These subjects will harbor cardiac sodium channel gene variants.
  Procainamide: One time intravenous infusion of Procainamide administered over 30 minutes. Dosage is calculated as 10mg/kg based on subject's ideal body weight.
Arm/Group | Atrial Fibrillation With ST Changes on Electrocardiogram
Number analyzed (Participants) | 89
Participants | 4
Statistical Analysis 1: Comparison: Atrial Fibrillation With ST Changes on Electrocardiogram; Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 0 — 0 participants with rare SCN5A non-synonymous variants met the primary outcome for ST-segment elevation; Given the very small number of outcomes (N=4) and the small number of participants with the primary determinant (N=2), a Fisher's Exact Test is the appropriate test and it yields a P-value=1.000

ADVERSE EVENTS:
Time Frame: 1 hour
Description: Adverse events definitions match ClinicalTrials.gov
Arm/Group | Atrial Fibrillation With ST Changes on Electrocardiogram
Serious Adverse Events (participants affected / at risk) | 1/106
Other Adverse Events (participants affected / at risk) | 6/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atrial Fibrillation With ST Changes on Electrocardiogram (N=106)
Cerebrovascular accident (CVA) post ablation (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atrial Fibrillation With ST Changes on Electrocardiogram (N=106)
Hypotension (Blood and lymphatic system disorders) | 1 (1)
Nause/Vomiting (Gastrointestinal disorders) | 4 (4)
Prolonged QT (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes